CLINICAL TRIAL: NCT04011657
Title: Effective Antimicrobial StewaRdship StrategIES (ARIES): Cluster-randomized Trial of a Computerized Decision Support System Versus Antibiotic Prospective Review and Feedback in Antimicrobial Stewardship
Brief Title: Effective Antimicrobial StewaRdship StrategIES (ARIES)
Acronym: ARIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015/00671
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Infection, Bacterial
Keywords: computerized decision support; prospective review and feedback; antimicrobial stewardship
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Masking Description: A parallel-group, 1:1 block-cluster randomized, cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voluntary CDSS (Experimental): Voluntary use of computerized decision support with prospective review and feedback
  Interventions: Other: Compulsory CDSS
- Compulsory CDSS (No Intervention): Compulsory use of computerized decision support with prospective review and feedback

INTERVENTIONS:
Other: Compulsory CDSS — Compulsory CDSS use with prospective review feedback in patients prescribed with piperacillin tazobactam or carbapenems
  Arms: Voluntary CDSS

SUMMARY:
Background Prospective review and feedback (PRF) of antibiotic prescriptions is a labor-intensive core strategy of antimicrobial stewardship (AMS). The investigators hypothesized that a computerized decision support system (CDSS) providing recommendations for antibiotics, investigations and referrals would reduce the requirement for PRF without causing harm.

Methods A parallel-group, 1:1 block-cluster randomized, cross-over study was conducted in 32 medical and surgical wards from March to August 2017. The intervention arm comprised voluntary use of CDSS at first prescription of piperacillin-tazobactam or a carbapenem, while the control arm was compulsory CDSS. PRF was continued for both arms. Primary outcome was 30-day mortality.

DETAILED DESCRIPTION:
Increasing antimicrobial resistance due to inappropriate antimicrobial use is a global concern. Multi-disciplinary antimicrobial stewardship teams have become an integral part of the response to this issue. Through prospective review of antibiotic prescriptions and feedback (PRF) to healthcare providers, antimicrobial stewardship has been shown to improve clinical response, reduce adverse effects and mortality. However, this strategy is labor-intensive to implement and skilled healthcare workers are an expensive and scarce resource. Antibiotic computerized decision support systems (CDSS) have been used to facilitate these processes and may circumvent the limitations of lack of manpower. In previous studies, CDSS led to increased susceptibility of Pseudomonas aeruginosa to imipenem and Enterobacteriaceae to gentamicin and ciprofloxacin, and an overall reduction in broad-spectrum antibiotic use. CDSS could improve clinical outcomes. Currently, there are limited studies comparing the combined effects of these two strategies.

At Tan Tock Seng Hospital, a university teaching hospital in Singapore, antimicrobial stewardship has focused on PRF by a multi-disciplinary team since 2009. This team reviews piperacillin-tazobactam and carbapenem orders against hospital antibiotic guidelines from day two of antibiotic prescription. In March 2010, we implemented CDSS triggered at the point of antibiotic ordering and compulsory for the prescriber to review. Prescribers are free to accept or reject the CDSS recommendations. While PRF and CDSS are performed following the same institutional guidelines, there may be differences in physicians' acceptance of recommendations and the accessibility to recommendations between these two interventions. In previous studies, PRF recommendations had an acceptance of 60-70% while compulsory CDSS was 40%. The investigators hypothesized that compulsory CDSS and PRF would improve clinical outcomes compared with voluntary CDSS and PRF, and compulsory CDSS would improve appropriate antibiotic practice and reduce the requirement for subsequent PRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are started on the 1st episode of piperacillin-tazobactam or carbapenem during the study period.
* Medical and surgical wards

Exclusion Criteria:

* Intensive care unit (ICU), high dependency and step-down care wards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
30-day mortality | Follow-up up to 30 days from the start date of the first episode of piperacillin-tazobactam or carbapenem use
  Death at 30 days

SECONDARY OUTCOMES:
7-day clinical response | Follow-up up to 7 days from the date of the first episode of piperacillin-tazobactam or carbapenem use
  resolution of systemic inflammatory response syndrome
30-day re-infection | Re-start of piperacilin-tazobactam or carbapenem 30 days after the cessation of first episode of piperacillin-tazobactam or carbapenem use
  Re-start of piperacilin-tazobactam or carbapenem 30 days after the cessation of first episode of piperacillin-tazobactam or carbapenem use
30-day readmission | Readmissions 30 days after the cessation of first episode of piperacillin-tazobactam or carbapenem use
  Readmission after the cessation of first episode of piperacillin-tazobactam or carbapenem use
length of stay | It is assessed from the date of admission till the date of discharge or up to 6 months
  Duration of admission
6-months incidence of multi-drug resistant organisms | up to 6 months (Clinical cultures only)
  MRSA, VRE, ESBL, MDR-A. baumannii, XDR- A baumannii, MDR- P. aeruginosa, XDR-P aeruginosa, C difficile , Carbapenem resistant enterobacterales
Diarrhea this admission | From the start date from the first episode of piperacillin-tazobactam or carbapenem use until the discharge date or up to 6 months whichever occurred earlier
  Incidence of diarrhea from start of first episode of piperacillin-tazobactam or carbapenem use till discharge
Appropriateness of antibiotics | It is assessed only once at the point of the first episode of piperacillin-tazobactam or carbapenem use in the index admission. It is only assessed once till discharge or up to 6 months
  first episode of piperacillin-tazobactam or carbapenem use according to hospital guidelines. Appropriateness will be described as "yes" or "no".
Index antibiotic days of therapy, | From the start date of the first episode of piperacillin-tazobactam or carbapenem use to the end date of this antibiotic which is followed up till discharge or up to 6 months.
  Duration of the first episode of piperacillin-tazobactam or carbapenem use
Gross hospitalization costs | Gross hospitalization costs incured from date of admission till date of discharge or up to 6 months
  Gross hospitalization costs

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be made available only after project agreement is made

REFERENCES:
- [Background] Barlam TF, Cosgrove SE, Abbo LM, MacDougall C, Schuetz AN, Septimus EJ, Srinivasan A, Dellit TH, Falck-Ytter YT, Fishman NO, Hamilton CW, Jenkins TC, Lipsett PA, Malani PN, May LS, Moran GJ, Neuhauser MM, Newland JG, Ohl CA, Samore MH, Seo SK, Trivedi KK. Implementing an Antibiotic Stewardship Program: Guidelines by the Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America. Clin Infect Dis. 2016 May 15;62(10):e51-77. doi: 10.1093/cid/ciw118. Epub 2016 Apr 13. PMID 27080992
- [Background] Davey P, Marwick CA, Scott CL, Charani E, McNeil K, Brown E, Gould IM, Ramsay CR, Michie S. Interventions to improve antibiotic prescribing practices for hospital inpatients. Cochrane Database Syst Rev. 2017 Feb 9;2(2):CD003543. doi: 10.1002/14651858.CD003543.pub4. PMID 28178770
- [Background] Lew KY, Ng TM, Tan M, Tan SH, Lew EL, Ling LM, Ang B, Lye D, Teng CB. Safety and clinical outcomes of carbapenem de-escalation as part of an antimicrobial stewardship programme in an ESBL-endemic setting. J Antimicrob Chemother. 2015 Apr;70(4):1219-25. doi: 10.1093/jac/dku479. Epub 2014 Dec 3. PMID 25473028
- [Background] Schuts EC, Hulscher MEJL, Mouton JW, Verduin CM, Stuart JWTC, Overdiek HWPM, van der Linden PD, Natsch S, Hertogh CMPM, Wolfs TFW, Schouten JA, Kullberg BJ, Prins JM. Current evidence on hospital antimicrobial stewardship objectives: a systematic review and meta-analysis. Lancet Infect Dis. 2016 Jul;16(7):847-856. doi: 10.1016/S1473-3099(16)00065-7. Epub 2016 Mar 3. PMID 26947617
- [Background] Yong MK, Buising KL, Cheng AC, Thursky KA. Improved susceptibility of Gram-negative bacteria in an intensive care unit following implementation of a computerized antibiotic decision support system. J Antimicrob Chemother. 2010 May;65(5):1062-9. doi: 10.1093/jac/dkq058. Epub 2010 Mar 9. PMID 20215130
- [Background] Thursky K. Use of computerized decision support systems to improve antibiotic prescribing. Expert Rev Anti Infect Ther. 2006 Jun;4(3):491-507. doi: 10.1586/14787210.4.3.491. PMID 16771625
- [Background] Leibovici L, Kariv G, Paul M. Long-term survival in patients included in a randomized controlled trial of TREAT, a decision support system for antibiotic treatment. J Antimicrob Chemother. 2013 Nov;68(11):2664-6. doi: 10.1093/jac/dkt222. Epub 2013 Jun 5. PMID 23743088
- [Background] Chow AL, Lye DC, Arah OA. Mortality Benefits of Antibiotic Computerised Decision Support System: Modifying Effects of Age. Sci Rep. 2015 Nov 30;5:17346. doi: 10.1038/srep17346. PMID 26617195